CLINICAL TRIAL: NCT06416930
Title: Study of Cadonilimab Combined With Chemotherapy in Recurrent / Refractory Pleural Mesothelioma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Akesobio (Industry)
Responsible Party: Principal Investigator, Jie Wang, Chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-039
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Pleural Mesothelioma
Keywords: Cadonilimab; pleural mesothelioma; Bispecific Antibody
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab combined with chemotherapy (Experimental): All subjects in the group will be treated with Cadonilimab plus gemcitabine / vinorelbine / pemetrexed once every three weeks.
  Interventions: Drug: Cadonilimab Combined with chemotherapy

INTERVENTIONS:
Drug: Cadonilimab Combined with chemotherapy — Cadonilimab (15mg/kg, intravenous drip, D1) + gemcitabine (1250mg/m2, intravenous drip, D1/D8) or vinorelbine (30mg, oral, tiw, D1/D3/D5) or pemetrexed (500mg/m2, intravenous drip, D1), every 3 weeks.
  Other Names: AK104

SUMMARY:
This is a multicenter, single-arm, phase II clinical study to evaluate the safety and efficacy of Cadonilimab combined with gemcitabine, or vinorelbine, or pemetrexed in the treatment of patients with recurrent / refractory pleural mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced or metastatic pleural mesothelioma;
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
3. Participants must have previously failed to receive platinum-containing chemotherapy with or without bevacizumab, and have received at most two-line systemic therapy.
4. Measurable disease as per mRECIST v1.1 for assessment of response in malignant pleural mesothelioma.
5. Adequate haematological, renal and liver function.

Exclusion Criteria:

1. Primary mesothelioma of peritoneum, pericardium and testes
2. Active, untreated central nervous system (CNS) metastasis.
3. Use of Chinese herbal medicine or immunomodulatory agents with anti-tumor indications within 14 days prior to the first dose of study treatment.
4. Known active autoimmune diseases.
5. Presence of other uncontrolled serious medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2027-06-20 (Estimated); Study Completion 2029-06-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 year
  defined as the percentage of participants who achieve a best overall response of complete response or partial response assessed according to mRECIST v1.1 for assessment of response in malignant pleural mesothelioma.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 2 year
  defined as the percentage of participants who achieve a best overall response of complete response, partial response, or stable disease assessed according to mRECIST v1.1 for assessment of response in malignant pleural mesothelioma.
Progression Free Survival (PFS) | 2 year
  defined as the time between the date of first dose of study drug and the date of first documented tumor progression per mRECIST v1.1, or death due to any cause, whichever occurs first.
Duration of Response (DoR) | 2 year
  defined as the interval from the date of first documentation of objective response (complete response or partial response, according to the mRECIST v1.1) to the date of first documented tumor progression, or death due to any cause, whichever occurs first.
Overall Survival (OS) | 2 year
  defined as the interval from the date of first documentation of objective response (complete response or partial response, according to the mRECIST v1.1) to the date of first documented tumor progression, or death due to any cause, whichever occurs first.
Adverse Events (AEs) | 2 year
  Incidence and severity of adverse events (AE) and clinically significant abnormal laboratory results